CLINICAL TRIAL: NCT05195385
Title: Lung Cancer Screening With Low-dose CT Scan in Women : Implementation Study
Acronym: CASCADE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministère de la Santé et des Solidarités (Unknown); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP210362; 2021-A02265-36 (Other: ID-RCB Number)
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer Screening
Keywords: lung neoplasms; multidetector computed tomography; early detection of cancer; artificial intelligence; lung cancer screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Procedure (Other): Baseline low dose Ct acquisition, then at 1 year and 2 years to depict suspicious lung nodules
  Interventions: Procedure: Low-dose computed tomography of the chest

INTERVENTIONS:
Procedure: Low-dose computed tomography of the chest — Baseline low dose Ct acquisition, then at 1 year and 2 years to depict suspicious lung nodules

SUMMARY:
The purpose of this study is to determine whether reading of low-dose thoracic CT scans can be done by a single general radiologist who has been trained to lung cancer screening, and will evaluate the performance in comparison with double reading by experts.

The study will enroll women between 50 and 74 years old, at risk for lung cancer due to their smoking history.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death, worldwide. Several randomized studies have demonstrated that annual or biennial low-dose CT screening reduces lung cancer mortality. However, these studies involved expert chest radiologists, with double reading being performed in most studies. Furthermore, none of the published studies have evaluated the role of artificial intelligence to serve as second of concurrent reader.

Women with at least 20 pack-year smoking history who quitted smoking less than 15 years ago will be enrolled to have baseline, 1-year and 2-year low-dose CT of the chest.

The CT scans will be read on site by a general radiologist trained to lung cancer screening according to the European lung cancer screening certification program, first without then with the aid of an artificial algorithm trained to lung nodule detection (Veye Chest, Aidence). All CT scans will also be read by 2 chest experts, who will resolve their disagreement by a consensus reading if necessary. Patient management will rely on the double reading by expert. The criteria for positive screen result are as follows: solid nodule > 500 mm3 (10 mm) or growing (30% volume increase), part-solid nodule with > 8 mm solid component or new or growing, pure ground glass nodule developing a solid portion.

ELIGIBILITY:
Inclusion Criteria:

* Women aged from 50 to 74 years
* who had smoked at least 20 pack years and quit less than 15 years ago
* Had given their consent and accepted the need for a 2-year follow-up
* Affiliated to the social security system

Exclusion Criteria

* Presence of clinical symptoms suggesting malignancy (weight loss, hemoptysis) or ongoing infection (cough with fever)
* Evolving cancer
* History of lung cancer
* A 2-year follow-up not possible
* Chest CT scan performed within 2 years prior to inclusion

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2635 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2027-10-08 (Estimated); Study Completion 2027-10-08 (Estimated)

PRIMARY OUTCOMES:
Performance of trained radiologists for lung cancer screening | 2 years
  Sensitivity, specificity, predictive values compared to double reading by experts

SECONDARY OUTCOMES:
Effectiveness of screening | 2 years
  Proportion of participants with a positive screening test and proportion of confirmed diagnosis of cancer
Analysis of the diagnostic performance of the reading without detection software, in order to assess its incremental value | 2 years
  For the general population and for the COPD population. Sensitivity, specificity, predictive values and likelihood ratios of the initial reading compared to the expert readings, using histological diagnosis as gold standard for positive screens and stability at 2 years for negative screens
Analysis of the performance of a reading by detection software alone | 2 years
  For the general population and for the COPD population. Sensitivity, specificity, predictive values and likelihood ratios of artificial intelligence alone
Analysis of the concordances of the different readings | 2 years
  Kappa concordance coefficient between the different readings
Adherence to screening | 2 years
  Number of participants related to the number of eligible women, having completed all the required scans (3 to 6), speed of inclusion in the study. Enrolment will be assessed on the basis of the following characteristics: weaned or non-weaned smokers, level of education, socio-economic category, etc
Analysis of the impact of screening on smoking cessation | 2 years
  Smoking cessation rate at the end of the study
Psychological impact of screening | 2 years
  HADS (Hospital Anxiety and Depression Scale) questionnaire at each scan, Cancer worry scale, Satisfaction with Decision scale at inclusion and end of study, all translated into French
Number of co-morbidities (COPD, coronary artery disease) detected | 2 years
  Number of participants related to the number of women included in the study for whom treatment is initiated (bronchodilators/ statins or revascularization/ osteoporosis treatment)
Evaluation of costs induced by screening | 2 years
  Cost measures: total cost of screening, average cost per woman, average cost per woman screened
Prevalence of osteoporosis by opportunistic screening | 2 years
  Presence of at least one thoracic vertebral fracture and measurement of trabecular attenuation of the T8 vertebral body

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre REVEL, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Marie WISLEZ, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôtel-Dieu, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Revel MP, Abdoul H, Chassagnon G, Canniff E, Durand-Zaleski I, Wislez M. Lung CAncer SCreening in French women using low-dose CT and Artificial intelligence for DEtection: the CASCADE study protocol. BMJ Open. 2022 Dec 8;12(12):e067263. doi: 10.1136/bmjopen-2022-067263. PMID 36600392